CLINICAL TRIAL: NCT06085989
Title: Nynnamm - Effects of Infant Directed Singing on Breastfeeding Difficulties
Acronym: Nynnamm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna University (Other)
Responsible Party: Principal Investigator, Jenny Ericson, Associated Professor, Dalarna University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 280958
Record Dates: First submitted 2023-06-16; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infant directed singing (Experimental): The intervention group will receive standard breastfeeding support from health care staff combined with maternal infant-directed singing during breastfeeding. The starting point of the singing will be individually assessed and tailored to the dyads and will start approximately a few minutes before breastfeeding starts. An educational video about how to apply infant-directed singing will be shown to all mothers in the intervention group.
  Interventions: Behavioral: Infant directed singing
- Standard care (Active Comparator): Mothers allocated to the control group will be offered standard breastfeeding support from health care staff, and data on secondary outcome measures will be collected during one breastfeeding session.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Infant directed singing — In every known human culture and historical period, infant-directed singing exists as a natural feature of parental care for newborn infants. Infant-directed singing is effective in regulating infant affect and in capturing an infant's attention for a longer period than infant-directed speech. Parental stress significantly decreases when parents are encouraged to use their own voices to soothe their infants with a song or a lullaby of their choice.
  Arms: Infant directed singing
Behavioral: Standard care — Standard breastfeeding support to mothers with breastfeeding difficulties provided by health care professionals.
  Arms: Standard care

SUMMARY:
Breastfeeding is one of the most effective, health economical interventions to promote health and reduce illness in both mothers and children. However, breastfeeding in Sweden is under threat. An increasing number of newborns will miss out on its benefits because lack of lactation support for mothers with breastfeeding difficulties, which is the main reasons for breastfeeding cessation. About 110,000 mothers breastfeed every year but the prevalence is decreasing. Many mothers are dissatisfied with the support they receive from health care. Maternal infant-directed singing could be an effective, person- and family-centered, cost-effective, self-care intervention to reduce stress and breastfeeding difficulties in new mothers as well as increasing oxytocin, which is an important hormone for lactation and well-being.

This project evaluates the effect of a self-care intervention involving maternal infant-directed singing during breastfeeding on maternal stress, experiences, and breastfeeding rates up to six months postpartum among mothers with breastfeeding difficulties. The mothers are randomized to standard care and infant-directed singing or control with standard care. The primary outcome is the proportion of breastfeeding four weeks after the intervention. 260 mothers will be included in the project, which will be conducted during 2024-2025, and data will be analyzed and presented in 2026. A data management plan will ensure that all research activities are well organized.

DETAILED DESCRIPTION:
In Sweden, there is an extensive restructuring of care in relation to the concept "good quality, local health care" (God och nära vård). Most new mothers are cared for at home in direct connection to birth, which places new demands on primary health care providers. A lack of knowledge and training for professionals will affect new mothers' opportunities to breastfeed to the extent that they wish. Furthermore, breastfeeding rates are decreasing in Sweden. Contributors to this trend could be health care-related factors, downsizing, staff shortages, and a lack of breastfeeding knowledge and supportive interventions. There is a risk for even lower breastfeeding rates when professionals lack supportive interventions for advising mothers. This is hazardous since its known that breastfeeding is an effective way to ensure child health and survival. Breastfeeding also provides significant health benefits for mothers and is a cost-effective way to reduce health care costs.

Purpose and aims The aim of this study is to evaluate the effect of a self-care intervention involving maternal infant-directed singing during breastfeeding on maternal stress, experiences, and breastfeeding rates up to six months postpartum among mothers with breastfeeding difficulties.

The specific aim of the study is to:

* investigate whether maternal infant-directed singing during breastfeeding is effective in increasing the breastfeeding rate 4 weeks after the intervention among mothers with breastfeeding difficulties (primary outcome).
* investigate whether maternal infant-directed singing during breastfeeding is effective in decreasing maternal stress and breastfeeding difficulties up to six months postpartum among mothers with breastfeeding difficulties (secondary outcome).
* describe maternal experiences of using infant-directed singing during breastfeeding among mothers who have breastfeeding difficulties (secondary outcome).
* investigate parent-infant moment-to-moment communication to provide a deeper understanding of breastfeeding situations and potential problems in this context (secondary outcome).
* investigate cortisol levels, sodium levels, and the somatic cell count in breast milk and saliva (cortisol only) among the participating mothers (secondary outcome).

Method Design An exploratory multicenter randomized controlled trial with two parallel groups with an allocation ratio of 1:1 is planned. The investigators hypothesize that a combination of standard breastfeeding support and maternal infant-directed singing during breastfeeding will improve the proportion of breastfeeding mothers, including the mother-infant dyad's experience, and decrease stress among mothers who have breastfeeding difficulties.

Participants and setting The study will be performed at different child health care centers and postnatal care facilities in the Dalarna, Uppsala and Värmland regions. Mothers who seek support for breastfeeding difficulties, including experiencing a low milk supply, sore nipples, and breast pain, feeling stressed or unwell while breastfeeding or having an infant who has problems with latching, will be eligible for inclusion. The participants must understand Swedish or English and be over 18 years old. During the health care visit, mothers will be informed about the study, and written informed consent will be obtained from the mothers who want to participate in the study.

Data collection and procedures The mothers will be randomized to one of two arms. The randomization will be performed by the health care staff or research team members using an automated and secure web-based system administered independently of the research team. Block randomization will be used, with blocks of 8 interventions and 8 controls.

The intervention group will receive standard breastfeeding support from health care staff combined with maternal infant-directed singing during breastfeeding. The starting point of the singing will be individually assessed and tailored to the dyads and will start approximately a few minutes before breastfeeding starts. An educational video about how to apply infant-directed singing will be shown to all mothers in the intervention group.

Mothers allocated to the control group will be offered standard breastfeeding support from health care staff, and data on secondary outcome measures will be collected during one breastfeeding session.

The health care staff will provide standard breastfeeding support to all mothers during their visit. Then, the mothers will breastfeed their infants. Before breastfeeding starts, the research team will collect baseline data (questions and biological samples) and connect the mothers to the Galvanic Skin Response (GSR) device, which measures changes in sweat gland activity that are reflective of the intensity of the mothers' emotional state/ arousal. The breastfeeding session will be video-recorded. After breastfeeding, the mothers will answer additional questions, and another saliva cortisol sample will be collected. The order may be different depending on infant hunger signals.

The research team will be available approximately 5-10 days a month during the data collection period, which is expected to last 1 ½ years.

Due to the nature of the intervention, blinding will not be possible for the health care staff and parents during the procedures. The research team will not be completely blinded; however, data collection will be performed by different researchers on different data collection days. Hence, no researcher will have full access to all mothers' randomization groups. The person calling to collect data for the primary outcome will be blinded. Additionally, for the secondary outcomes, the research team will be blinded to a large extent.

Data analysis and statistics A priori power analysis will be used to examine the power necessary to detect an 11% difference between the two groups in the breastfeeding prevalence 4 weeks after the intervention. There is a need to include 121 mothers in the intervention group and 121 mothers in the control group to be able to reject the null hypothesis that the proportion of breastfeeding mothers in the intervention and control groups is equal with a probability (power) of 0.8 using logistic regression. To account for possible dropouts, an additional 18 (nine in each group) mothers will be recruited, leaving us with a total sample of 260 mother-infant dyads. The Type I error probability associated with this test of the null hypothesis is 0.05.

An intention-to-treat approach will be used during the analysis. To analyze the data, several statistical models and qualitative methods will be used. The primary outcome-breastfeeding (yes/no)-will be analyzed with logistic regression analysis presented with odds ratios and 95% confidence intervals. Depending on the distribution of the variables, the secondary outcomes will be analyzed with appropriate comparative statistical models. Quantitative data will also be presented using descriptive statistics. Qualitative data (i.e., open-ended questions, notes, comments, interview data) will be analyzed with a qualitative content analysis. The video recordings and singing will be analyzed with microanalysis. Microanalysis can be defined as a social microscope, an in-depth, hand-coded, second-by-second analysis method of video footage, which may provide a deeper understanding of breastfeeding situations and potential problems in this context. With microanalysis, the investigators will, for example, be able to discern synchronicity and timing or the lack thereof in breastfeeding mothers on a micro level, providing research with knowledge on a macro level on how to better guide mothers in similar situations. Mixed methods will be used when analyzing data. Quantitative and qualitative data will first be analyzed separately and thereafter merged and interpreted as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who seek support for breastfeeding difficulties.
* Mothers who seek support for experiencing a low milk supply.
* Mothers who seek support for sore nipples.
* Mothers who seek support for breast pain.
* Mothers who seek support for feeling stressed.
* Mothers who seek support for feeling unwell while breastfeeding.
* Mothers who seek support for having an infant who has problems with latching the breast.
* Must understand Swedish or English.
* Must be over 18 years old.

Exclusion Criteria:

* Living outside Region Dalarna, Sweden
* Living outside Region Uppsala, Sweden
* Living outside Region Värmland, Sweden

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 260 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of breastfeeding (yes/no) four weeks after the intervention assessed by telephone | 4 weeks after health care visit (intervention)
  The primary outcome is the proportion of breastfeeding (yes/no) mothers 4 weeks after the intervention, and data on the primary outcome will be collected by telephone by a research nurse.

SECONDARY OUTCOMES:
Maternal stress assessed by galvanic skin response (GSR), area small peaks, which is obtained via three electrodes on the maternal palm. | Two minutes before, after three minutes breastfeeding and two minutes after the breastfeeding session at the intervention visit
  Mothers' emotional state/ arousal (stress) before, during and after the breastfeeding session, measured with the GSR device.
Maternal stress assessed by galvanic skin response (GSR) area huge peaks, which is obtained via three electrodes on the maternal palm. | Two minutes before, after three minutes breastfeeding and two minutes after the breastfeeding session at the intervention visit
  Mothers' emotional state/ arousal (stress) before, during and after the breastfeeding session, measured with the GSR device.
Maternal stress assessed by galvanic skin response (GSR), peaks per second, which is obtained via three electrodes on the maternal palm. | Two minutes before, after three minutes breastfeeding and two minutes after the breastfeeding session at the intervention visit
  Mothers' emotional state/ arousal (stress) before, during and after the breastfeeding session, measured with the GSR device.
Maternal stress assessed by galvanic skin response (GSR), average rise time, which is obtained via three electrodes on the maternal palm. | Two minutes before, after three minutes breastfeeding and two minutes after the breastfeeding session at the intervention visit
  Mothers' emotional state/ arousal (stress) before, during and after the breastfeeding session, measured with the GSR device.
Maternal stress assessed by galvanic skin response (GSR), average peak, which is obtained via three electrodes on the maternal palm. | Two minutes before, after three minutes breastfeeding and two minutes after the breastfeeding session at the intervention visit
  Mothers' emotional state/ arousal (stress) before, during and after the breastfeeding session, measured with the GSR device.
Proportion of breastfeeding (yes/no) at 2 and 4 weeks after the intervention and at 2, 4, 6 months of infant age. | Two and 4 weeks after intervention, 2, 4, 6 months of infant age.
  The proportion of breastfeeding mothers 2 weeks after the health care visit and when the infant is 2, 4 and 6 months of age. These data will be collected by telephone by a research nurse.
Breastfeeding status assessed by five questions about latch, suction power and pattern, maternal feeling and nipple shape. | Before intervention, 2 and 4 weeks after intervention, 2, 4, 6 months of infant age.
  Breastfeeding status (five questions) will be determined before the intervention. Additionally, these questions will be asked at 2 and 4 weeks after the intervention and at 2, 4 and 6 months of age by telephone.
  Higher scores indicate greater problems. Latch scored 1-5 Pain while breastfeeding, scored 1-4 Suction power, scored 1-4 Suction pattern, scored 1-3 Nipple shape, scored 1-4 Minimum 5 points and maximum 20 points
Biological samples of breast milk to determine the somatic cell count. | During health care visit (intervention) on day 1
  Samples will be collected during the health care visit to determine the somatic cell count (cells per milliliter) in breast milk.
Biological samples of breast milk to determine the sodium levels. | During health care visit (intervention) on day 1
  Samples will be collected during the health care visit to determine the sodium levels in mmol/L.
Biological samples of saliva and hair to determine cortisol levels in the mother and infant. | During health care visit (intervention) on day 1
  Samples will be collected during the health care visit to determine the saliva cortisol levels (mothers and infants), and hair cortisol levels (mothers only).
Maternal experience of infant directed singing and breastfeeding support they received during the health care visit assessed by a qualitative interviews about four weeks after the intervention. | Four weeks after the intervention
  Semistructured interviews (with 25 mothers in the intervention group) will be conducted about the experiences of using infant-directed singing in connection to breastfeeding.
Maternal experience of infant directed singing and breastfeeding support they received during the health care visit assessed by yes/no, likert scale and open ended questions in a survey sent home to the mothers about four weeks after the intervention. | Four weeks after the intervention
  Maternal experiences of using infant-directed singing in connection to breastfeeding. The mothers will be asked a few questions about the intervention and breastfeeding support in a survey sent home to the mothers 4 weeks after the intervention.
  Likert scale maximum 5 and minimum 1, higher scores indicate higher satisfaction with singing and support.
Micro analysis assessed by a qualitative video observation of multi modal interaction activities by the mother and infant (verbal and non-verbal interactions). | During the breastfeeding session at the health care visit (intervention) on day 1
  Video recordings will be taken during the intervention for the microanalysis of the breastfeeding session, breastfeeding positions and breastfeeding combined with mother's infant-directed singing.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Ericson, Docent, Principal Investigator — Dalarna University

IPD SHARING:
Plan to Share IPD: No
Can not be shared due to ethical regulations.